CLINICAL TRIAL: NCT06995482
Title: A Phase 1, Open Label, Randomized, Multiple Ascending Dose (MAD) Study Evaluating the Safety, Tolerability and Pharmacokinetics of KSHN001034 in Healthy Postmenopausal Female Volunteers
Brief Title: Multiple Ascending Dose Study to Evaluate the Safety, Tolerability and Pharmacokinetics of KSHN001034 in Healthy Postmenopausal Female Volunteers
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Kashiv BioSciences, LLC (Industry)
Collaborators: Eric Solutions LLC (Unknown); Clinexcel Research, Ahmedabad, India (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: CE-24-06
Record Dates: First submitted 2025-05-19; First posted 2025-05-29 (Actual); Last update posted 2026-02-12 (Actual); Status verified 2026-02

CONDITIONS: Healthy Postmenopausal Women
MeSH Terms: interventions — Fulvestrant

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (5):
- Cohort 1 (Experimental)
  Interventions: Drug: KSHN001034; Drug: Fulvestrant
- Cohort 2 (Experimental)
  Interventions: Drug: KSHN001034; Drug: Fulvestrant
- Cohort 3 (Experimental)
  Interventions: Drug: KSHN001034; Drug: Fulvestrant
- Cohort 4 (Experimental)
  Interventions: Drug: KSHN001034; Drug: Fulvestrant
- Cohort 5 (Experimental)
  Interventions: Drug: KSHN001034; Drug: Fulvestrant

INTERVENTIONS:
Drug: KSHN001034 — Test Product: KSHN001034, 5 mL vial containing 113 mg/mL of KSHN001034, equivalent to 100 mg/mL of fulvestrant. Manufactured for Kashiv Biosciences LLC, USA.
  • 6 subjects will receive low dose of KSHN001034 IM on Days 1, 8, 15, and 22.
  Arms: Cohort 1
Drug: KSHN001034 — Test Product: KSHN001034, 5 mL vial containing 113 mg/mL of KSHN001034, equivalent to 100 mg/mL of fulvestrant. Manufactured for Kashiv Biosciences LLC, USA.
  • 6 subjects will receive medium dose of KSHN001034 IM on Days 1, 8, 15, and 22.
  Arms: Cohort 2
Drug: KSHN001034 — Test Product: KSHN001034, 5 mL vial containing 113 mg/mL of KSHN001034, equivalent to 100 mg/mL of fulvestrant. Manufactured for Kashiv Biosciences LLC, USA.
  • 6 subjects will receive high dose of KSHN001034 IM on Days 1, 8, 15, and 22.
  Arms: Cohort 3
Drug: KSHN001034 — Test Product: KSHN001034, 5 mL vial containing 113 mg/mL of KSHN001034, equivalent to 100 mg/mL of fulvestrant. Manufactured for Kashiv Biosciences LLC, USA.
  • 6 subjects will receive low dose of KSHN001034 SC on Days 1, 8, 15, and 22.
  Arms: Cohort 4
Drug: KSHN001034 — Test Product: KSHN001034, 5 mL vial containing 113 mg/mL of KSHN001034, equivalent to 100 mg/mL of fulvestrant. Manufactured for Kashiv Biosciences LLC, USA.
  • 6 subjects will receive medium dose of KSHN001034 SC on Days 1, 8, 15, and 22.
  Arms: Cohort 5
Drug: Fulvestrant — Reference Product: Faslodex® (Fulvestrant), 5 mL pre-filled syringe containing 250 mg/5 mL of fulvestrant, administered as two 5 mL injections (total 500 mg) via intramuscular (IM) injection. Marketed by AstraZeneca.
  • 2 subjects will receive 500 mg Fulvestrant IM on Days 1 and 15.

SUMMARY:
The goal of this clinical trial is to evaluate if KSHN001034 demonstrates safety, tolerability, and a comparable pharmacokinetic (PK) profile to the reference product, Faslodex® (fulvestrant), which is used for the treatment of hormone receptor-positive breast cancer.

Participants will:

Receive either the test product (KSHN001034) or the reference product (Faslodex®) administered intramuscularly (IM) or subcutaneously (SC) at doses of low, medium, or high , with doses conducted in 5 cohorts and these participants will be healthy postmenopausal female volunteers.

Dosing will be administered in a sequential cohort-wise manner across five cohorts, with DSMB oversight for safety monitoring and dose escalation.

Primary Endpoint:

Safety and tolerability will be assessed based on the occurrence, severity, and relationship of adverse events (AEs), including serious adverse events (SAEs).

Secondary Endpoint:

Pharmacokinetic (PK) parameters will be evaluated, including Cmax (maximum concentration), Tmax (time to maximum concentration), AUC (area under the curve), and T1/2 (half-life).

DETAILED DESCRIPTION:
A phase 1, Open Label, Randomized, Multiple Ascending Dose (MAD) study to evaluate the safety, tolerability, and pharmacokinetics (PK) of KSHN001034 in comparison with US-licensed Faslodex® (Fulvestrant) administered through intramuscular (IM) and subcutaneous (SC) routes in healthy postmenopausal female volunteers. Participants will be randomized in a 3:1 ratio to receive either KSHN001034 (administered IM or SC at low, medium, or high dose in five cohorts) or the reference product, Faslodex® (500 mg IM). Dose escalation will proceed cohort-wise, based on DSMB review of cumulative safety and PK data. PK blood samples will be collected from Day 1 to Day 36 across multiple pre- and post-dose timepoints to estimate PK parameters. Safety assessments include adverse events (AEs), serious adverse events (SAEs) as assessed by CTCAE v5.0.

ELIGIBILITY:
Inclusion Criteria:

1. Able to provide written Informed Consent and communicate with the investigator and comprehend study-related procedures.
2. Healthy, postmenopausal females aged 45 to 60 years old (inclusive), as determined by medical history and physical examination.
3. Body Mass Index at screening between 18 and 30 kg/m2, inclusive.
4. Post-menopausal females (Menopause is defined as the female is either 12 months off menstrual period after the age of 50 years, or 12 months off menstrual period after the age of 45 years and FSH > 40 mIU/mL Note: Amenorrhea should not be due to lactation).
5. Participant must be healthy on the basis of their medical history, a physical examination, vital signs, and 12-lead Electrocardiogram (ECG) performed during screening and as determined by the Principal Investigator (PI).
6. Hemoglobin at screening and Day (-1) ≥ 11 g/dl
7. Ability to communicate well and to comply with the requirements of the entire study.
8. Adequate venous access and can able to give required blood samples.

Exclusion Criteria:

1. History or presence of cardiovascular, pulmonary, hepatic, renal, hematologic, coagulation, gastrointestinal, endocrine, immunologic, dermatologic, neurologic, or psychiatric disease or any other clinical significant abnormalities during screening investigations which, in the opinion of the PI, may either put the participant at risk because of participation in the study, or influence the results or the participant's ability to participate in the study.
2. Evidence of organ dysfunction [e.g. liver dysfunction; ≥ Upper Limit of Normal (ULN) for ALT, AST or ALP or renal dysfunction (<90 mL/min of creatinine clearance by Cockroft-Gault formula] or any clinically significant abnormalities in other clinical laboratory parameters at screening as determined by the investigator.
3. QTc (Bazzett) interval ≥450 ms on ECG at screening.
4. Any major surgery requiring general anesthesia within 3 months prior to screening.
5. Known or suspected history of alcohol dependency or addictive substance use, as judged by the investigator Note: Participants will be required to abstain from recreational use of soft addictive substances (such as marijuana) within 2 weeks or hard addictive substances (such as cocaine, phencyclidine, crack, opioid derivatives including heroin, and amphetamine derivatives) within 2 months prior to screening
6. History or presence of malignancy in the last 5 years
7. Positive testing for human immunodeficiency virus (HIV I or II), hepatitis B (hepatitis B surface antigen [HBsAg]), or hepatitis C (Anti-HCV antibody) at screening.
8. Received or intending to receive a vaccination in the two weeks prior to dosing, or anytime during study participation.
9. Donated blood within 60 days of screening or otherwise experienced blood loss of >250 mL within the same period.
10. Presence of low platelet count (i.e. lower than LLN), bleeding issues or family history of bleeding disorders.
11. Participant has a history of hypersensitivity to heparin as checked at screening.
12. History of hypersensitivity or idiosyncratic reaction to test drug or any drug chemically similar to the drug under investigation or any of the excipients.
13. The participant has any estrogen- dependent conditions including benign breast conditions
14. The participant has a history of osteoporosis or any disease affecting bone or steroid metabolism.
15. Intolerance to/ fear of venipuncture, needles, or blood draws.
16. Positive serum pregnancy test during screening or Lactating mothers
17. Has received another new chemical entity/investigational drug within 28 days or 5 half-lives of investigational drug (whichever is longer) of the first administration of investigational product in this study.
18. Use of any prescribed or non-prescribed medication, herbal remedies, megadose vitamins (intake of 20 to 600 times the recommended daily dose) and minerals during the 2 weeks prior to the first administration of investigational product.
19. The participant has consumed grapefruit-containing beverages and foods 7 days prior to dosing.
20. Any condition that, in the opinion of the investigator, might interfere with study objectives.
21. Subjects with abnormal international normalized ratio (INR) at screening

Ages: 45 Years to 60 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes
Enrollment: 40 (Estimated)
Dates: Start 2025-08-18 (Actual); Primary Completion 2026-05 (Estimated); Study Completion 2026-06 (Estimated)

PRIMARY OUTCOMES:
Number of participants with treatment-related Adverse events as assessed by CTCAE v5.0 | up to 36 days after dosing
  Adverse events reported after dosing will be evaluated

SECONDARY OUTCOMES:
Pharmacokinetic parameter | upto day 36 after dosing
  Evaluate the Peak Plasma Concentration (Cmax)
Pharmacokinetic parameter | upto day 36 after dosing
  Evaluate the Area under the plasma concentration versus time curve (AUC)
Pharmacokinetic parameter | up to 36 days after dosing
  Evaluate the Time to maximum concentration (Tmax)
Pharmacokinetic parameter | up to 36 days after dosing
  Evaluate the half life (T1/2)

CONTACTS AND LOCATIONS:
Locations (2):
- Floridian Clinical Research LLC, Miami Lakes, Florida, United States
- Synergen Bio Pvt. Ltd., Pune, Maharashtra, India